CLINICAL TRIAL: NCT02450383
Title: Comparison of Two Different Surgical Approaches to Increase Peri-Implant Mucosa Thickness: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Two Different Surgical Approaches To Increase Peri-Implant Mucosa Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Gustavo Avila-Ortiz, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201407810
Record Dates: First submitted 2015-01-26; First posted 2015-05-21 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Tooth Loss; Peri-implant Mucosa Defect
MeSH Terms: conditions — Tooth Loss | interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Autologous subepithelial connective tissue graft
  Interventions: Procedure: Autologous subepithelial connective tissue graft
- Experimental (Experimental): Acellular Dermal Matrix
  Interventions: Drug: Acellular Dermal Matrix

INTERVENTIONS:
Drug: Acellular Dermal Matrix — Placement of acellular dermal matrix (Alloderm®) on the buccal/coronal aspect of the alveolar ridge at the time of implant placement, following a two-stage approach
  Other Names: Alloderm®
  Arms: Experimental
Procedure: Autologous subepithelial connective tissue graft — Placement of autologous subepithelial connective tissue graft on the buccal/coronal aspect of the alveolar ridge at the time of implant placement, following a two-stage approach
  Other Names: sCTG
  Arms: Control

SUMMARY:
The purpose of this non-inferiority trial is to determine the clinical efficacy of acellular dermal matrix (ADM) in the augmentation of the gum around dental implants as compared to an autologous gum graft (sCTG) obtained from the palate (roof of the mouth) in human adults.

AlloDerm is regulated by the US Food and Drug Administration (FDA) as human tissue for transplantation. AlloDerm is processed and marketed in accordance with the FDA's requirements for banked human tissue (21 CFR, Part 1270 and Part 1271) and Standards for Tissue Banking of the American Association of Tissue Banks (AATB).

Twenty adult subjects will be recruited who are in need of dental implant placement with simultaneous gum grafting to increase the thickness of the facial mucosa. Half of the subjects will be randomized to the ADM group and half will be randomized to the sCTG group. The surgical intervention will be performed according to the protocol and subjects will return for follow-up 2, 4, 8, and 16 weeks post-surgery for follow-up measurements of healing, gum thickness, subject perception of pain, and esthetic photographs.

DETAILED DESCRIPTION:
Although little is known about the influence of peri-implant mucosa thickness (PMT) on long-term biologic outcomes, soft tissue thickness is a critical component to esthetic dental implant restorations. While the subepithelial connective tissue graft (sCTG) has been recognized as the gold standard for gingival augmentation, several studies have reported acellular dermal matrix (ADM) may produce similar outcomes. Healthy patients with a thin biotype were selected on the basis of an eligibility criteria and randomized to the control (sCTG) or test (ADM) group. Measurements were completed by a masked examiner at baseline and at implant uncovering. Patient reported outcomes were recorded, as well. A power analysis suggested 20 subjects be recruited. The gain in PMT at 1mm, 3mm and 5mm from the expected CEJ and recipient site wound dehiscence were measured and recorded in both groups at different time points by a calibrated, masked examiner. Patient-related outcome measures (PROMs), such as pain and level of satisfaction with final outcome, were also recorded for all study participants.

ELIGIBILITY:
Inclusion criteria:

* Age: 18 to 80 years.
* Subjects must be able and willing to follow instructions related to the study procedures.
* Subjects must have read, understood and signed an informed consent form.
* At least one single-tooth edentulous site, with adjacent natural teeth, planned for tooth replacement therapy with an implant-supported restoration.

Exclusion criteria:

* Reported allergy or hypersensitivity to any of the products to be used in the study.
* Severe hematologic disorders, such as hemophilia or leukemia.
* Active severe infectious diseases that may compromise normal healing.
* Liver or kidney dysfunction/failure.
* Currently under cancer treatment or within 18 months from completion of radio- or chemotherapy.
* Subjects with uncontrolled diabetes, defined as Hba1c > 6.5% (According to the American Diabetes Association 2014 Guidelines)
* Pregnant women or nursing mothers.
* Smokers: Subjects who have smoked within 6 months of study onset.
* Concomitant medications for systemic conditions that may affect the outcomes of the study.
* Any other non-specified reason that from the point of view of the investigators will make a candidate not a suitable subject for the study (e.g. limited mouth opening).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Avila-Ortiz, DDS, MS, PhD, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa College of Dentistry - Craniofacial Clinical Research Center and Department of Periodontics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning on sharing IPD

REFERENCES:
- [Derived] Hutton CG, Johnson GK, Barwacz CA, Allareddy V, Avila-Ortiz G. Comparison of two different surgical approaches to increase peri-implant mucosal thickness: A randomized controlled clinical trial. J Periodontol. 2018 Jul;89(7):807-814. doi: 10.1002/JPER.17-0597. Epub 2018 Jul 20. PMID 29633268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in January 2015 and was finalized in May 2016
Groups:
- Control: Implant placement with subepithelial connective tissue graft
  Autologous subepithelial connective tissue graft
- Experimental: Implant placement with simultaneous acellular dermal matrix graft (human allograft)
  Alloderm®
Period: Overall Study
Arm/Group | Control | Experimental
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.0) | 59.7 (10.9) | 55.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Peri-implant mucosa thickness at 1 mm [Mean (Standard Deviation); unit: millimeters] | 3.05 (1.28) | 2.85 (1.40) | 3.0 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Buccal Peri-implant Mucosa Thickness Between Baseline and 16 Weeks After Surgery
Description: Buccal mucosa thickness measurements were obtained by a calibrated, masked examiner using a custom-made stent and an endo file for precision and reproducibility between different time points
Time Frame: Baseline and 16 weeks after baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 10
millimeters | 0.44 (2.04) | 0.05 (1.57)

2. Secondary Outcome: Changes in Peri-implant Keratinized Mucosa Width (Apico-coronal) at 16 Weeks After Surgery
Time Frame: Baseline to 16 weeks after baseline
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 10
millimeters | -0.85 (1.13) | -0.45 (1.30)

3. Secondary Outcome: Patient-perceived Discomfort, Measured by VAS
Description: Patient-reported outcome measures of perceived discomfort using a visual analog scale (VAS) from 0 (no pain) to 100 (maximum pain) were recorded
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 10
units on a scale | 23.60 (24.71) | 10.10 (7.78)

4. Secondary Outcome: Wound Healing, Measured Using a Standardized Visual Wound Healing Index
Description: Wound healing status was evaluated by the same calibrated clinician using a standardized visual wound healing index at different time points A simple wound healing scoring system including 3 categories was used: 1- uneventful wound healing, 2- slight gingival edema, erythema or discomfort, 3- poor wound healing
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 10 | 10
units on a scale | 1.70 (0.48) | 1.90 (0.57)

ADVERSE EVENTS:
Time Frame: Baseline intervention to 16 weeks after baseline
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | Experimental (N=10)
Early Wound Dehiscence (Surgical and medical procedures) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes